CLINICAL TRIAL: NCT01611454
Title: Prospective Randomized Evaluation of a New Fabric Attenuation Device in Endovascular Interventional Radiology II (PREFER II)
Brief Title: New Fabric Attenuation Device in Endovascular Interventional Radiology II (PREFER II)
Acronym: PREFER-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Principal Investigator, Raul Herrera, MD, Director, Division of Clinical Research & Outcomes, Baptist Health South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PREFER II
Record Dates: First submitted 2012-05-02; First posted 2012-06-05 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Occupational Exposure to Radiation
Keywords: Occupational Exposure to Radiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XPF thyroid collar (Experimental): Administration of the XPF Thyroid Collar during the same type of interventional radiology procedures as Comparator arm above
  Interventions: Device: XPF thyroid collar
- Equivalent collar (Active Comparator): Administration of the Standard 0.5mm lead-equivalent thyroid collar during the same type of interventional radiology procedures as Comparator arm above.
  Interventions: Device: Standard 0.5mm lead equivalent thyroid collar

INTERVENTIONS:
Device: XPF thyroid collar — Interventionalist wear the experimental (XPF) thyroid collar during fluoroscopy guided interventions.
  Arms: XPF thyroid collar
Device: Standard 0.5mm lead equivalent thyroid collar — Interventionalist wear a standard 0.5mm lead equivalent thyroid collar during the same type of comparator fluoroscopy guided interventions. Comparator arm uses same type of lead thyroid collar but the XPF under investigation.
  Arms: Equivalent collar

SUMMARY:
The PREFER II trial primary objective of the trial is to show how much radiation attenuation is provided by XPF thyroid collars in absolute and relative terms.

DETAILED DESCRIPTION:
The PREFER II trial has three main objectives. The primary objective of the trial is to show how much radiation attenuation is provided by XPF thyroid collars in absolute and relative terms. The secondary objective of the study is to measure and compare the amount of radiation that interventional radiologists are exposed to per case in an interventional suite setting using FDA approved XPF thyroid collars or standard 0.5 mm Pb equivalent thyroid collars.

The third objective is to assess the operator comfort wearing the XPF protection devices. In order to achieve these objectives, measurements will be performed in 150 consecutive interventional procedures requiring C-arm fluoroscopy performed at BCVI. A prospective randomization will be performed, assigning participants to wear their own standard 0.5 mm Pb equivalent thyroid collar or to wear the FDA approved XPF thyroid collar. Radiation exposure will be monitored with 2 radiation detectors (TLDs, one inside and one outside the thyroid collar) which the participant is required to wear. After each procedure the participant will be asked to rate the comfort of wearing the devices on a scale from 1 to 100.

ELIGIBILITY:
Inclusion Criteria:

* Interventional Radiologists practicing in Baptist Cardiac & Vascular Institute
* consecutive endovascular procedure requiring C-arm fluoroscopy

Exclusion Criteria:

* Interventional Neuroradiologists and Interventional Cardiologists will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry T Katzen, MD, Principal Investigator — Baptist Hospital of Miami, Baptist Cardiac and Vascular Institute; Heiko Uthoff, MD, Principal Investigator — Baptist Hospital of Miami, Baptist Cardiac and Vascular Institute
Locations (1):
- Baptist Hospital of Miami, Baptist Cardiac and Vascular Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rowe VL, Lee W, Weaver FA, Etzioni D. Patterns of treatment for peripheral arterial disease in the United States: 1996-2005. J Vasc Surg. 2009 Apr;49(4):910-7. doi: 10.1016/j.jvs.2008.11.054. PMID 19341885

RESULTS

PARTICIPANT FLOW:
Groups:
- XPF Thyroid Collar: Administration of the XPF Thyroid Collar.
  XPF thyroid collar: Interventionalist wear the experimental (XPF) thyroid collar during fluoroscopy guided interventions.
- Equivalent Collar: Administration of the Standard 0.5mm lead-equivalent thyroid collar.
  Standard 0.5mm lead equivalent thyroid collar: Interventionalist wear a standard 0.5mm lead equivalent thyroid collar during fluoroscopy guided interventions.
Period: Overall Study
Arm/Group | XPF Thyroid Collar | Equivalent Collar
Started | 58 | 48
Completed | 40 | 38
Not Completed | 18 | 10
Not completed — Lack of Efficacy | 18 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XPF Thyroid Collar | Equivalent Collar | Total
Number analyzed (Participants) | 58 | 48 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 26 | 62
  >=65 years | 22 | 22 | 44
Age, Continuous [Median (Standard Deviation); unit: Year] | 50 (25) | 50 (25) | 50 (25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 32 | 24 | 56
Region of Enrollment [Number; unit: participants]
  United States | 58 | 48 | 106

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change
Description: Radiation attenuation. The null hypothesis is that the XPF thyroid collar is equal to the standard 0.5mm Pb lead equivalent thyroid collar with regard to radiation attenuation/transmission in relative (%) terms. The alternative hypothesis is that the XPF thyroid collar is superior or inferior to the standard thyroid collar. Based on our results obtained during the 60 procedures (PREFER trial), 150 procedures are required to demonstrate a significant difference with an alpha level of 5% and a power of 80%. Radiation attenuation percentage is measure by interrogation of the lead attenuates X-rays counter required to be used in all interventional radiology clinical procedures by each physician operator. The interrogation is done by measuring the energy imparted per unit mass in the counter wore by ionizing radiation to matter at the specified point. The International System of Units (SI) unit of absorbed dose is the joule per kilogram.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | XPF Thyroid Collar | Equivalent Collar
Number analyzed (Participants) | 58 | 48
percentage change | 79.7 (25.8) | 71.9 (34.2)

2. Secondary Outcome: Wearing Comfort of the Collar on a Scale From 0-100.
Description: Operators are asked directly after each procedure to rate the wearing comfort, graded worst to best. 0 means low comfort (worse outcome) and 100 is the best comfort level (best outcome) with wearing the collar.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | XPF Thyroid Collar | Equivalent Collar
Number analyzed (Participants) | 58 | 48
score on a scale | 85.0 (8.8) | 83.3 (13.1)

3. Secondary Outcome: Radiation Exposure (uSv) for for Both the Thyroid and Equivalent Collars
Description: (day 1) Operators are asked directly after each procedure to rate the wearing comfort Radiation exposure will be monitored with radiation detectors (TLDs, 2 attached to the collar) which the participant is required to wear. Exposure is measured as the energy imparted per unit mass by ionizing radiation to the matter at the specified time of the procedure. The International System of Units (SI) unit of absorbed dose is the joule per kilogram. The special name for this unit is the gray (Gy). For purposes of radiation protection and assessing dose or risk to humans in general terms, the quantity normally calculated is the mean absorbed dose in an organ or tissue.
Time Frame: 1 day
Population: XPF thyroid collar and the equivalent collar are combined under one outcome measure as the outcome measure is comparing the arms and not as individual measures.
Measure: Mean (Standard Deviation); unit: Gy
Groups:
- Dose Measured Outside Collar; Dose Measured Inside Collar: Radiation exposure will be monitored with radiation detectors, which the participant is required to wear. It will be measured based on uSv's.
Arm/Group | Dose Measured Outside Collar | Dose Measured Inside Collar
Number analyzed (Participants) | 106 | 106
Gy | 272.3 (373.3) | 98.2 (203.1)

4. Secondary Outcome: Radiation Exposure (uSv) for XPF Caps and the Equivalent Caps
Description: (day 1) Operators are asked directly after each procedure to rate the wearing comfort Radiation exposure will be monitored with radiation detectors, which the participant is required to wear. Exposure is measured as the energy imparted per unit mass by ionizing radiation to the matter at the specified time of the procedure. The International System of Units (SI) unit of absorbed dose is the joule per kilogram. The special name for this unit is the gray (Gy). For purposes of radiation protection and assessing dose or risk to humans in general terms, the quantity normally calculated is the mean absorbed dose in an organ or tissue.
Time Frame: 1 day
Population: XPF caps and the equivalent caps are combined under one outcome measure as the outcome measure is comparing the arms and not as individual measures.
Measure: Mean (Standard Deviation); unit: Gy
Groups:
- Dose Measured Outside Cap: Radiation exposure will be monitored with radiation detectors outside the cap, which the participant is required to wear. It will be measured based on uSv's.
- Dose Measured Inside Cap: Radiation exposure will be monitored with radiation detectors inside the cap, which the participant is required to wear. It will be measured based on uSv's.
Arm/Group | Dose Measured Outside Cap | Dose Measured Inside Cap
Number analyzed (Participants) | 106 | 106
Gy | 224.1 (266.1) | 48.1 (124.7)

ADVERSE EVENTS:
Arm/Group | XPF Thyroid Collar | Equivalent Collar
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/48
Other Adverse Events (participants affected / at risk) | 0/58 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No